CLINICAL TRIAL: NCT01574456
Title: Blood-brain Barrier Permeability in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL36156.068.11
Record Dates: First submitted 2012-04-05; First posted 2012-04-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- 7 patients diagnosed with dementia of the Alzheimer's type
- 13 patients with mild cognitive impairment
- 19 healthy controls

SUMMARY:
The main aim of the present study is to improve our understanding of the role of blood-brain barrier function in dementia of the Alzheimer's type. The investigators hypothesize that microvascular dysfunction - more specifically "cerebral perfusion and blood-brain barrier leakage" - is a determinant of cognitive decline and cortical atrophy in Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

Patients with AD:

* Informed consent before participation in the study
* Received standard diagnostic procedure according to the Parelsnoer Initiative procedure
* Diagnosed with dementia of the Alzheimer's type
* Clinical dementia rating (CDR) of 1, which means a mild to moderate stage of dementia
* MMSE ≥ 20 and patients are mentally competent (in general, individuals with an MMSE ≥ 18 are considered mentally competent)

Patients with prodromal AD:

* Informed consent before participation in the study
* Received standard diagnostic procedure according to the Parelsnoer Initiative procedure
* Diagnosis of prodromal dementia according to the Dubois criteria (16)
* CDR of 0.5, which suggests a very mild stage of dementia
* Memory impairment defined as Delayed Recall on Verbal Learning Test (15 WLT) < 1.5 SD
* MMSE ≥ 20 and patients are mentally competent.
* Medial temporal lobe atrophy scale MTA ≥ 1 (17) OR abnormal levels of Aß42, t-tau or p-tau

Healthy participants:

* Informed consent before participation in the study
* No Diagnosis of dementia, prodromal dementia, or mild cognitive impairment.
* MMSE ≥ 26
* No substantial memory complaints (according to participant)
* Age, gender and education is matched to the patient groups.

Exclusion Criteria:

* Contraindications for scanning (e.g. brain surgery, cardiac pacemaker, metal implants, claustrophobia, large body tattoos)
* Contraindications for contrast agent Gadovist (renal failure) as determined by the estimated Glomular Filtration Rate eGFR < 30 mL/min.
* Major vascular disorders (e.g. stroke, heart disease)
* Psychiatric or neurological disorders: Major depression (< 12 months); history of schizophrenia; bipolar disorder; psychotic disorder NOS or treatment for a psychotic disorder (< 12 mnd); cognitive impairment due to alcohol abuse; epilepsy; Parkinson's disease; MS; brain surgery; brain trauma; electroshock therapy; kidney dialysis; Meniere's disease; and brain infections.
* Structural abnormalities of the brain
* Cognitive impairment due to alcohol/drug abuse
* Absence of reliable informant (for patient groups)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three groups of participants have been included: 7 patients diagnosed with dementia of the Alzheimer's type; 13 patients with mild cognitive impairment due to AD, which represents a preclinical stage of AD in which patients already have memory impairment and at least one AD biomarker (i.e. hippocampal atrophy or abnormal amyloid and tau protein content in the cerebrospinal fluid); and 19 healthy controls. Patients have been recruited from the memory clinics of the Maastricht University Medical Center and the Leiden University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The main study measures are blood brain barrier permeability as measured by T1-weighted dynamic contrast MRI | 22 months

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Leids University Medical Center, Leiden
  - Maastricht University Hospital, Maastricht